CLINICAL TRIAL: NCT03617081
Title: A First Human Dose Trial Investigating the Safety, Tolerability and Pharmacokinetics of Single Doses of Oral NNC0113-2023 in Healthy Male Subjects
Brief Title: First Research Study of the Possible New Medicine NNC0113-2023 in Healthy Men.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9023-4408; U1111-1209-3837 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-08-01; First posted 2018-08-06 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC0113-2023 (Experimental): Participants will receive increasing doses of NNC0113-2023 on day 1. Each participant will receive only a single dose.
  Interventions: Drug: NNC0113-2023
- Placebo (Placebo Comparator): Participants will receive placebo (NNC0113-2023)
  Interventions: Drug: Placebo (NNC0113-2023)

INTERVENTIONS:
Drug: NNC0113-2023 — Participants will receive dose levels of 1 mg, 2 mg, 4 mg, 8 mg, 16 mg or 32 mg of NNC0113-2023 orally. Each participant will receive only one dose.
  Arms: NNC0113-2023
Drug: Placebo (NNC0113-2023) — Participants will receive NNC0174-0833 matched placebo orally.
  Arms: Placebo

SUMMARY:
The aim of this study is to assess how safe the study drug is and how well a participant tolerates it after a single oral (taken by mouth) dose. The study also aims to measure the concentration of the study drug and its breakdown products after a single dose. Participants will either get NNC0113-2023 (a new medicine) or placebo (a "dummy medicine similar to the study medicine but without active ingredients) - which treatment any participant gets is decided by chance. Participants will get one dose (can be one or two tablets) of study medicine. The study will last for about 65 days. Participants will have 10 scheduled site visits with the study physician or study staff at the study centre. For one of the visits, participants will stay at the research unit for 5 days. At all visits, except the first information visit, participants will have blood drawn along with other clinical assessments. Participants cannot take part in this study if participants have any disorder that the doctor thinks is a health problem. Only healthy men are allowed to take part.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 - 45 years (both inclusive) at the time of signing informed consent.
* Body mass index between 20.0 kg/m^2 and 29.9 kg/m^2 (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* HbA1c greater than or equal to 6.5 % (48 mmol/mol) at screening.
* Use of tobacco and nicotine products, defined as any of the below: 1) Smoking more than 1 cigarettes or the equivalent per day or 2) Not willing to refrain from smoking and use of nicotine substitute products during the in-house period.
* History of major surgical procedures involving the stomach potentially affecting absorption of trial products (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).
* Presence of clinically significant gastrointestinal disorders or symptoms of gastrointestinal disorders potentially affecting absorption of drugs or nutrients, as judged by the investigator.
* Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma.
* Presence or history of pancreatitis (acute or chronic).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From time of dosing (day 1) until completion of the follow-up visit (day 43)
  Count of events

SECONDARY OUTCOMES:
AUC0-∞,2023,SD; the area under the NNC0113-2023 plasma concentration-time curve from time 0 to infinity after a single dose of oral NNC0113-2023 | From baseline (day 1) to post treatment follow-up (day 43)
  Measured in nmol/L*h
Cmax,2023,SD; the maximum plasma concentration of NNC0113-2023 after a single dose of oral NNC0113-2023 | From baseline (day 1) to post treatment follow-up (day 43)
  Measured in nmol/L
AUC0-24h,SNAC,SD; the area under the SNAC plasma concentration-time curve from time 0 to 24 hours after a single dose of oral NNC0113-2023 | From baseline (day 1) to 24 hours after dosing
  Measured in ng/mL*h
Cmax,SNAC,SD; the maximum plasma concentration of SNAC in plasma after a single dose of oral NNC0113-2023 | From baseline (day 1) to 24 hours after dosing
  Measured in ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com